CLINICAL TRIAL: NCT04158466
Title: A Study to Evaluate the Safety and Efficacy of a Kalifilcon A Contact Lens for Daily Disposable Use
Brief Title: A Study to Evaluate the Safety and Efficacy of Kalifilcon A Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 890
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Contact Lens Wear
Keywords: Disposable Contact Lenses; Soft Contact Lens; Soft Contact Lenses

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Kalifilcon A Daily Disposable Contact Lenses (Experimental): Participants will wear Bausch + Lomb kalifilcon A daily disposable contact lenses for at least 8 hours per day at least 5 days per week for approximately 3 months. Participants will be provided with Bausch + Lomb Sensitive Eyes Drops for use as needed during the study and lens cases for return of worn study lenses to the Investigator at the end of the study.
  Interventions: Device: Kalifilcon A Daily Disposable Contact Lenses
- Biotrue ONEday Daily Disposable Contact Lenses (Active Comparator): Participants will wear Bausch + Lomb Biotrue ONEday daily disposable contact lenses for at least 8 hours per day at least 5 days per week for approximately 3 months. Participants will be provided with Bausch + Lomb Sensitive Eyes Drops for use as needed during the study and lens cases for return of worn study lenses to the Investigator at the end of the study.
  Interventions: Device: Biotrue ONEday Daily Disposable Contact Lenses

INTERVENTIONS:
Device: Kalifilcon A Daily Disposable Contact Lenses — Contact lens
  Arms: Kalifilcon A Daily Disposable Contact Lenses
Device: Biotrue ONEday Daily Disposable Contact Lenses — Contact lens
  Other Names: Bausch + Lomb Biotrue ONEday® Daily Contact Lens
  Arms: Biotrue ONEday Daily Disposable Contact Lenses

SUMMARY:
This study is to evaluate the safety and efficacy of a new silicone hydrogel daily disposable contact lens, kalifilcon A compared to the Bausch + Lomb Biotrue ONE day® daily disposable contact lens when worn by current soft contact lens wearers on a daily disposable wear basis.

DETAILED DESCRIPTION:
Approximately 247 participants (494 eyes) will be enrolled in at approximately 20 investigative sites in the United States (US). A minimum of 20% of the randomized participants will be of Japanese descent (for example, both maternal and paternal grandparents born in Japan).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.
* Participants must be myopic and require lens correction from -0.25 to -6.00 Diopter (D) with 0.25 D steps, in each eye.
* Participants must be correctable through spherocylindrical refraction and with soft spherical contact lenses to 40 letters (0.14 logMAR) or better (2 meters distance, high-contrast chart) in each eye.
* Participants must be free of any anterior segment disorders.
* Participants must be adapted soft contact lens wearers and willing to wear their study lenses for at least 8 hours per day at least 5 days per week on a daily disposable wear basis for approximately 3 months.
* Participants must be willing and able to comply with all treatment and follow-up/study procedures, as well as willing and able to refrain from using any other contact lenses or solutions other than those provided for the duration of the study.

Exclusion Criteria:

* Participation in any drug or device clinical investigation within 2 weeks prior to entry into this study (Screening/Dispensing Visit) and/or during the period of study participation.
* Participants who are women of childbearing potential (those who are not surgically sterilized or postmenopausal) are excluded from participation in the investigation if they are currently pregnant, plans to become pregnant during the study, or is breastfeeding
* Participants who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last 3 months.
* Participants with any systemic disease currently affecting ocular health or in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Participants using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Participants with an active ocular disease or who are using any ocular medication.
* Participants who currently wear monovision, multifocal, or toric contact lenses.
* Participants with an ocular astigmatism of greater than 1.00 D in either eye.
* Participants with anisometropia (spherical equivalent) of greater than 2.00 D.
* Participants with any Grade 2 or greater finding during the slit lamp examination. Participants with corneal infiltrates of any grade.
* Participants with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Participants with any scar or neovascularization within the central 6 millimeters (mm) of the cornea.
* Participants who are aphakic.
* Participants who are amblyopic.
* Participants who have had any corneal surgery (for example, refractive surgery).
* Participants who are allergic to any component in the study care products.
* The participant is an employee of the investigative site.
* The participant, or a member of the participant's household, is an Ophthalmologist, an Optometrist, an Optician, or an Ophthalmic Assistant/Technician.
* The participant, or a member of the participant's household, is an employee of a manufacturer of contact lenses or contact lens care products (for example, Alcon, Bausch + Lomb, Ciba Vision, CooperVision, Johnson & Johnson).
* The participant, or a member of the participant's household, is an employee of a market research firm.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Donatello, Study Director — Bausch & Lomb Incorporated
Locations (16):
- United States (16):
  - Bausch Site 8, Los Angeles, California
  - Bausch Site 9, San Francisco, California
  - Bausch Site 10, Torrance, California
  - Bausch Site 12, Torrance, California
  - Bausch Site 6, Sarasota, Florida
  - Bausch Site 16, Honolulu, Hawaii
  - Bausch Site 4, ‘Aiea, Hawaii
  - Bausch Site 7, Pittsburg, Kansas
  - Bausch Site 11, Bloomington, Minnesota
  - Bausch Site 1, St Louis, Missouri
  - Bausch Site 13, Vestal, New York
  - Bausch Site 2, State College, Pennsylvania
  - Bausch Site 14, Brentwood, Tennessee
  - Bausch Site 5, Memphis, Tennessee
  - Bausch Site 3, Nashville, Tennessee
  - Bausch Site 15, New Berlin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 252 participants randomized but 251 participants received treatment. Participants are summarized by actual treatment group received.
Period: Overall Study
Arm/Group | Kalifilcon A Daily Disposable Contact Lenses | Biotrue ONEday Daily Disposable Contact Lenses
Started | 124 | 127
Completed | 121 | 126
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants are summarized by actual treatment group received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kalifilcon A Daily Disposable Contact Lenses | Biotrue ONEday Daily Disposable Contact Lenses | Total
Number analyzed (Participants) | 124 | 127 | 251
Age, Continuous [Mean (Full Range); unit: years] | 35.9 [18 to 54] | 33.6 [18 to 55] | 34.7 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 182
  Male | 36 | 33 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 60 | 55 | 115
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 59 | 64 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Average Daily Wear Time [Mean (Full Range); unit: hours per day] | 13.5 [8 to 18] | 13.4 [8 to 24] | 13.4 [8 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Mean logMAR Contact Lens Visual Acuity
Description: Visual acuity (VA) will be reported as letters read correctly, and the letters read will be converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant will read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters will be recorded. A decrease in the number of correct letters indicates a decrease in visual acuity. Acuity will be averaged across visits.
Time Frame: 3 months
Population: The per protocol population consisted of randomized without important (major) protocol deviations. It is a subset of the participants randomized and treated.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Kalifilcon A Daily Disposable Contact Lenses | Biotrue ONEday Daily Disposable Contact Lenses
Number analyzed (Participants) | 120 | 127
Number analyzed (eyes) | 240 | 254
units on a scale | -0.066 (0.0034) | -0.060 (0.0032)

2. Primary Outcome: Proportion of Participants With Slit Lamp Findings Greater Than Grade 2
Description: During an examination of both eyes without lenses, graded slit lamp findings will be assessed for each eye using Grades 0 (none), 1 (trace), 2 (mild), 3 (moderate), and 4 (severe). Using only the non-missing observations from all visits without imputation, each eye will be classified with respect to findings greater than Grade 2 at any visit (Absent or Present). Epithelial edema, epithelial microcysts, corneal staining, limbal Injection, bulbar injection, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates will be evaluated.
Time Frame: 3 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Kalifilcon A Daily Disposable Contact Lenses | Biotrue ONEday Daily Disposable Contact Lenses
Number analyzed (Participants) | 124 | 127
Number analyzed (eyes) | 248 | 254
eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were not coded, therefore source vocabulary is not applicable.
Arm/Group | Kalifilcon A Daily Disposable Contact Lenses | Biotrue ONEday Daily Disposable Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/127
Other Adverse Events (participants affected / at risk) | 0/124 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04158466/Prot_SAP_000.pdf